CLINICAL TRIAL: NCT05652296
Title: Post-Market Clinical Follow-up Registry of the Integra External Ventricular Drainage Systems and Accessories
Brief Title: External Ventricular Drainage Post-Market Clinical Follow-up Registry
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: C-EXTVDR-001
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cerebrospinal; Disorder
MeSH Terms: conditions — Central Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: External Ventricular Drainage (EVD) — EVD of Cerebral Spinal Fluid from the lateral ventricles of the brain

SUMMARY:
This post-market follow-up registry will capture clinical data specific to the safety and performance of the Integra External Ventricular Drainage Systems and Accessories.

DETAILED DESCRIPTION:
The purpose of this study is to investigate whether the Integra External Ventricular Drainage System listed as part of this study do perform to clinical expectations.

Additionally, this study will focus on the safety of these devices by collecting any device-specific Adverse Events (AEs) or Device deficiencies (DDs) seen when used during standard of care procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patient and/or legally authorized representative has agreed to participate in the study by signing the EC-approved consent form, where applicable.
2. Patients (of any age) who underwent or who plan to have a procedure with one of the Integra or Codman External Ventricular Drainage System.
3. For patients who have had the EVD System removed prior to study enrollment, have available follow-up data from implant until the EVD System is no longer required for drainage and monitoring of CSF.

Exclusion Criteria:

1. The Patients in whom more than one EVD System were or are intended to be placed.
2. The Patient has sepsis.
3. The Patient has a history of poor wound healing.
4. The patient exhibits signs of scalp infection prior to implantation that would be contraindicated per the IFU.
5. The Patient is otherwise determined by the Investigator to be medically unsuitable for participation in this Registry.
6. The Patient is currently enrolled in another device trial or has been previously entered in this trial.
7. The Patient is a prisoner or member of a different vulnerable population that should not be included in the study per the investigator.
8. The Patients known to have uncorrected coagulopathy.
9. The Patients with known hypersensitivity to rifampin or clindamycin hydrochloride (prior to implantation of Bactiseal catheters)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients of any age, and gender who underwent a procedure with one of the Integra External Ventricular Drainage Systems or Accessories
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Marzuola, Study Director — Integra LifeSciences Corporation
Locations (4):
- Belgium (3):
  - Ziekenhuis Oost-limburg, Genk
  - University Hospitals leuven, Leuven
  - AZ Delta, Roeselare
- Hôpital Gui de Chauliac, Montpellier, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive subjects of any age, and gender who gave consent for study participation, and who met the eligibility criteria and, who underwent a procedure with one of the Integra External Ventricular Drainage Systems or Accessories were enrolled into the study. The enrollment occured at at four sites in EU: three in Belgium and one in France.
Pre-assignment Details: A total of 120 patients, ie, the full consecutive series of patients from study sites were screened, and 117 subjects were included in this study.
Groups:
- Subject Underwent a Procedure With One Integra External Ventricular Drainage System or Accessorie.: Consecutive subjects of any age, and gender who gave consent for study participation, and who met the eligibility criteria and, who underwent a procedure with one of the Integra External Ventricular Drainage Systems or Accessories were enrolled into the study. The enrollment occured at at four sites in EU: three in Belgium and one in France. A total of 120 patients, ie, the full consecutive series of patients from study sites were screened, and 117 subjects were included in this study.
Period: Overall Study
Arm/Group | Subject Underwent a Procedure With One Integra External Ventricular Drainage System or Accessorie.
Started | 117
Completed | 104
Not Completed | 13

BASELINE CHARACTERISTICS:
Population: Subject Underwent a Procedure With one of the Integra External Ventricular Drainage Systems or Accessories.
Arm/Group | Subject Underwent a Procedure With One Integra External Ventricular Drainage System or Accessorie.
Number analyzed (Participants) | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (18.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 79
  France | 38

OUTCOME MEASURES:

1. Primary Outcome: Anticipated Drainage of Cerebrospinal Fluid (CSF)
Description: Percentage of subjects with anticipated drainage (i.e., observed drainage consistent with the patient's clinical presentation) of cerebrospinal fluid (CSF) in the clinical setting until the EVD System is no longer required.
Time Frame: 1 month following device implantation
Population: Subject underwent a procedure with one of the Integra External Ventricular Drainage Systems or Accessories.
Measure: Count of Participants; unit: Participants
Arm/Group | Subject Underwent a Procedure With One Integra External Ventricular Drainage System or Accessorie.
Number analyzed (Participants) | 117
Participants | 116

2. Secondary Outcome: Success of the Access to the Intracranial Space
Description: Percentage of subjects in whom the CODMAN Cranial Access Kit, when used with appropriate accessories, provided successful access to the intracranial space.
Time Frame: 1 month following device implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Subject Underwent a Procedure With One Integra External Ventricular Drainage System or Accessorie.
Number analyzed (Participants) | 117
Participants | 0

3. Other Pre Specified Outcome: Device- or Procedure Related Adverse Events (AEs) During the Use of the Device in the Patient
Description: Percentage of subjects with device related adverse events (AEs) during the use of the device in the patient
Time Frame: 1 month following device implantation
Population: Subject underwent a procedure with one of the Integra External Ventricular Drainage Systems or Accessories.
Measure: Count of Participants; unit: Participants
Arm/Group | Subject Underwent a Procedure With One Integra External Ventricular Drainage System or Accessorie.
Number analyzed (Participants) | 117
Participants | 81

4. Other Pre Specified Outcome: Noted Device Deficiencies During Use of the Device Such as Malfunction, Use Errors, or Other Issues Related to the Performance or Safety of the External Ventricular Drainage Systems and Accessories
Description: Percentage of subjects with noted Device Deficiencies during use of the device such as malfunction, use errors, or other issues related to the performance or safety of the External Ventricular Drainage Systems and Accessories
Time Frame: 1 month following device implantation
Population: Subject underwent a procedure with one of the Integra External Ventricular Drainage Systems or Accessories.
Measure: Count of Participants; unit: Participants
Arm/Group | Subject Underwent a Procedure With One Integra External Ventricular Drainage System or Accessorie.
Number analyzed (Participants) | 117
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse Event information were collected on any adverse event that the subject experienced within 1 month following device implantation.
Arm/Group | Subject Underwent a Procedure With One Integra External Ventricular Drainage System or Accessorie.
All-Cause Mortality (participants affected / at risk) | 10/117
Serious Adverse Events (participants affected / at risk) | 59/117
Other Adverse Events (participants affected / at risk) | 54/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subject Underwent a Procedure With One Integra External Ventricular Drainage System or Accessorie. (N=117)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 3 (4)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Brain death (General disorders) | 1 (1)
Condition aggravated (General disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Oedema (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (3)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2)
Bacterial infection (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
CNS ventriculitis (Infections and infestations) | 5 (5)
Device related sepsis (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3)
Postoperative wound infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1)
Unintentional medical device removal (Injury, poisoning and procedural complications) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1)
Bacterial test positive (Investigations) | 2 (2)
CSF cell count increased (Investigations) | 1 (1)
CSF volume increased (Investigations) | 1 (1)
Cerebral salt-wasting syndrome (Metabolism and nutrition disorders) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Cerebellar haematoma (Nervous system disorders) | 1 (1)
Cerebral vasoconstriction (Nervous system disorders) | 2 (2)
Cerebrospinal fluid leakage (Nervous system disorders) | 6 (8)
Epilepsy (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (5)
Hydrocephalus (Nervous system disorders) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 6 (7)
Loss of consciousness (Nervous system disorders) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1)
Device dislocation (Product Issues) | 2 (2)
Device leakage (Product Issues) | 1 (1)
Device occlusion (Product Issues) | 7 (8)
Product contamination (Product Issues) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 18 (20)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Wound drainage (Surgical and medical procedures) | 1 (1)
Surgery (Surgical and medical procedures) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1)
Vasospasm (Vascular disorders) | 12 (12)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subject Underwent a Procedure With One Integra External Ventricular Drainage System or Accessorie. (N=117)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Ear swelling (Ear and labyrinth disorders) | 1 (1)
Haematotympanum (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 4 (5)
Hypothyroidism (Endocrine disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (12)
Vomiting (Gastrointestinal disorders) | 5 (8)
Asthenia (General disorders) | 1 (1)
Complication associated with device (General disorders) | 2 (2)
Fatigue (General disorders) | 3 (3)
Pyrexia (General disorders) | 14 (17)
Bacteraemia (Infections and infestations) | 1 (1)
CNS ventriculitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Nosocomial infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Pneumonia aspiration (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebral ventricle dilatation (Nervous system disorders) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 7 (7)
Cognitive disorder (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 15 (24)
Intracranial pressure increased (Nervous system disorders) | 2 (2)
Partial seizures (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 4 (4)
Status epilepticus (Nervous system disorders) | 1 (1)
Subdural hygroma (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Device dislocation (Product Issues) | 1 (1)
Device occlusion (Product Issues) | 2 (2)
Product contamination (Product Issues) | 2 (2)
Agitation (Psychiatric disorders) | 2 (2)
Confusional state (Psychiatric disorders) | 2 (2)
Disorientation (Psychiatric disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Vasospasm (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-07-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT05652296/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT05652296/SAP_001.pdf